CLINICAL TRIAL: NCT01707134
Title: An Open-labelled, Controlled, Multicentre, Multinational, Extension Study Assessing Safety and Efficacy of the Human Insulin Analogue Insulin Aspart (X14) and Human Soluble Insulin as Meal Related Insulin in a Multiple Injection Regimen in Type 1 Diabetic Subjects
Brief Title: Safety and Efficacy of Insulin Aspart in Subjects With Type 1 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ANA/DCD/050
Record Dates: First submitted 2012-10-10; First posted 2012-10-16 (Estimated); Last update posted 2017-01-04 (Estimated); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1 | interventions — Insulin Aspart; Insulin, Isophane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- insulin aspart (Experimental)
  Interventions: Drug: insulin aspart; Drug: insulin NPH
- human insulin (Active Comparator)
  Interventions: Drug: human soluble insulin; Drug: insulin NPH

INTERVENTIONS:
Drug: insulin aspart — Injected subcutaneously (s.c, under the skin) as meal time insulin
  Arms: insulin aspart
Drug: human soluble insulin — Injected subcutaneously (s.c, under the skin) as meal time insulin
  Arms: human insulin
Drug: insulin NPH — Will be administrated subcutaneously (s.c, under the skin) once or twice daily as basal insulin

SUMMARY:
This trial is conducted in Europe. The aim of this trial is to evaluate the safety profile of insulin aspart in subjects with type 1 diabetes having participated in trial ANA/DCD/035.

ELIGIBILITY:
Inclusion Criteria:

* The subject must have completed the six month controlled treatment period in trial ANA/DCD/035

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 753 (Actual)
Dates: Start 1997-09; Primary Completion 2000-05 (Actual); Study Completion 2000-05 (Actual)

PRIMARY OUTCOMES:
Number of hypoglycaemic events

SECONDARY OUTCOMES:
Occurrence of adverse events
Incidence of hypoglycaemic episodes
Standard safety parameters: Haematology and biochemistry
HbA1c (glycosylated haemoglobin)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR,1452), Study Director — Novo Nordisk A/S
Locations (74):
- Austria (2):
  - Novo Nordisk Investigational Site, Graz
  - Novo Nordisk Investigational Site, Vienna
- Denmark (5):
  - Novo Nordisk Investigational Site, Copenhagen
  - Novo Nordisk Investigational Site, Frederiksberg
  - Novo Nordisk Investigational Site, Gentofte Municipality
  - Novo Nordisk Investigational Site, Kolding
  - Novo Nordisk Investigational Site, Køge
- Finland (4):
  - Novo Nordisk Investigational Site, Helsinki
  - Novo Nordisk Investigational Site, Kotka
  - Novo Nordisk Investigational Site, Kuopio
  - Novo Nordisk Investigational Site, Vantaa
- Germany (24):
  - Novo Nordisk Investigational Site, Bad Neuenahr-Ahrweiler
  - Novo Nordisk Investigational Site, Bad Oeynhausen
  - Novo Nordisk Investigational Site, Bochum
  - Novo Nordisk Investigational Site, Essen
  - Novo Nordisk Investigational Site, Flensburg
  - Novo Nordisk Investigational Site, Frankfurt
  - Novo Nordisk Investigational Site, Freiburg im Breisgau
  - Novo Nordisk Investigational Site, Friedrichsthal
  - Novo Nordisk Investigational Site, Giessen
  - Novo Nordisk Investigational Site, Haan
  - Novo Nordisk Investigational Site, Hamburg
  - Novo Nordisk Investigational Site, Kiel
  - Novo Nordisk Investigational Site, Magdeburg
  - Novo Nordisk Investigational Site, Mainz
  - Novo Nordisk Investigational Site, Mönchengladbach
  - Novo Nordisk Investigational Site, München
  - Novo Nordisk Investigational Site, Oberhausen
  - Novo Nordisk Investigational Site, Ostercappeln
  - Novo Nordisk Investigational Site, Saarlouis
  - Novo Nordisk Investigational Site, Schwerin
  - Novo Nordisk Investigational Site, Stuttgart
  - Novo Nordisk Investigational Site, Wiesbaden
  - Novo Nordisk Investigational Site, Wuppertal
  - Novo Nordisk Investigational Site, Würzburg
- Norway (5):
  - Novo Nordisk Investigational Site, Bergen
  - Novo Nordisk Investigational Site, Haugesund
  - Novo Nordisk Investigational Site, Oslo
  - Novo Nordisk Investigational Site, Stavanger
  - Novo Nordisk Investigational Site, Trondheim
- Sweden (2):
  - Novo Nordisk Investigational Site, Falun
  - Novo Nordisk Investigational Site, Karlstad
- Novo Nordisk Investigational Site, Zurich, Switzerland
- United Kingdom (31):
  - Novo Nordisk Investigational Site, Airdrie
  - Novo Nordisk Investigational Site, Bath
  - Novo Nordisk Investigational Site, Blackburn
  - Novo Nordisk Investigational Site, Bolton
  - Novo Nordisk Investigational Site, Church Village
  - Novo Nordisk Investigational Site, Cosham
  - Novo Nordisk Investigational Site, Coventry
  - Novo Nordisk Investigational Site, Edinburgh
  - Novo Nordisk Investigational Site, Exeter
  - Novo Nordisk Investigational Site, Gillingham
  - Novo Nordisk Investigational Site, Hull
  - Novo Nordisk Investigational Site, Inverness
  - Novo Nordisk Investigational Site, Leicester
  - Novo Nordisk Investigational Site, London
  - Novo Nordisk Investigational Site, Middlesbrough
  - Novo Nordisk Investigational Site, Newcastle
  - Novo Nordisk Investigational Site, Northampton
  - Novo Nordisk Investigational Site, Nottingham
  - Novo Nordisk Investigational Site, Penarth
  - Novo Nordisk Investigational Site, Plymouth
  - Novo Nordisk Investigational Site, Reading
  - Novo Nordisk Investigational Site, Rugby
  - Novo Nordisk Investigational Site, Salisbury
  - Novo Nordisk Investigational Site, Sheffield
  - Novo Nordisk Investigational Site, Southampton
  - Novo Nordisk Investigational Site, Stevenage
  - Novo Nordisk Investigational Site, Stirling
  - Novo Nordisk Investigational Site, Swansea
  - Novo Nordisk Investigational Site, Watford
  - Novo Nordisk Investigational Site, Whiston
  - Novo Nordisk Investigational Site, York

REFERENCES:
- [Result] Home PD, Hallgren P, Usadel KH, Sane T, Faber J, Grill V, Friberg HH. Pre-meal insulin aspart compared with pre-meal soluble human insulin in type 1 diabetes. Diabetes Res Clin Pract. 2006 Feb;71(2):131-9. doi: 10.1016/j.diabres.2005.05.015. Epub 2005 Jul 27. PMID 16054266
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com